CLINICAL TRIAL: NCT02636621
Title: Efficacy of Oral Appliance for Upper Airway Resistance Syndrome: Randomized, Parallel, Placebo, Controlled Study
Brief Title: Efficacy of Oral Appliance for Upper Airway Resistance Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Sonia Maria Guimaraes Pereira Togeiro Moura, Prof. Dra. Sonia Guimaraes Togeiro Moura, Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SR94036
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Upper Airway Resistance Syndrome
Keywords: Fatigue; excessive daytime sleepiness; flow limitation
MeSH Terms: conditions — Fatigue; Disorders of Excessive Somnolence | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brazilian Dental Appliance (Active Comparator): The device increases the volume of the airway by mandibular traction.
  Interventions: Device: Brazilian Dental Appliance
- Placebo (Placebo Comparator): Oral device that does not change the volume of the airway
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Brazilian Dental Appliance — Brazilian Dental Appliance is an oral appliance worn only during sleep that supports the jaw in a forward position to help maintain an open upper airway.
  Other Names: Mandibular advancement device
  Arms: Brazilian Dental Appliance
Other: Placebo — The placebo consists in a protective dental plate worn only during sleep that do not interfere in the size of the upper airway.
  Other Names: Protective dental plate
  Arms: Placebo

SUMMARY:
Introduction: The Upper Airway Resistance Syndrome (UARS) is a sleep disorder characterized by airway resistance to breathing during sleep that leads to arousals and daytime sleepiness. There are few studies about UARS treatment and there is not any gold standard treatment for it yet.

Objective: Primary: To evaluate the efficacy of oral appliance on improving fatigue in patients with UARS. Secondary: Evaluate the effects of treatment with oral appliance (OA) in patients with UARS on sleepiness, mood, cognition, quality of life, metabolism and autonomic nervous system.

Methods: Subjects with UARS (Apnea/Hypopnea Index - AHI - ≤ 5 events per hour of sleep and Respiratory Disturbance Index - RDI - > 5 events per hour or more than 30% of total sleep time with inspiratory flow limitation and with excessive daytime somnolence and/or fatigue) of both genders, with body mass index (BMI) lower than 30Kg/m2 and between 25 to 50 years of age will be included. Subjects will be randomly distributed in OA group and placebo (without treatment). At baseline evaluation, 6 months and 1 year after subjects will be submitted to sleep questionnaires, physical exam, otolaryngological evaluation, baseline polysomnography, Epworth sleepiness scale, Multiple Sleep Latency Test, fatigue scale, neurocognitive testing, autonomic nervous system analysis (heart rate variability) and metabolic evaluation. Mean and standard deviation will be used for descriptive statistical analysis if normal distribution, and median and percentiles (25%, 75%) for variables not normally distributed. To compare treatment groups T test (parametric) and Mann Whitney (non parametric) will be used. For adjusted analysis, linear regression analysis will be used.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Body mass index (BMI) ≤ 30Kg/m2
* Age from 25 to 50 years
* Clinical and polysomnographic diagnosis of Upper Airway Resistance Syndrome: Apnea/Hypopnea Index (AIH) ≤ 5 events/hour and Respiratory Disturbance Index (RDI) > 5 events/hour or > 30% of total sleep time with inspiratory flow limitation with excessive daytime somnolence or fatigue

Exclusion Criteria:

* Unsatisfactory dental condition or severe temporomandibular disfunction;
* Nasal obstruction;
* Alcohol abuse and excessive consumption of psychotropic drugs;
* Clinical, neurological or psychiatric diseases not treated
* Less than 6 hours of sleep

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Fatigue | From the baseline evaluation to one year after the treatment with oral appliance
  Modified fatigue impact scale for Portuguese (MFIS- BR)

SECONDARY OUTCOMES:
Subjective excessive daytime sleepiness | From the baseline evaluation to one year after the treatment with oral appliance
  Epworth sleepiness scale
Objective excessive daytime sleepiness | From the baseline evaluation to one year after the treatment with oral appliance
  Multiple Sleep Latency Test
Mood - Anxiety | From the baseline evaluation to one year after the treatment with oral appliance
  Beck inventories (BAI)
Mood - Depression | From the baseline evaluation to one year after the treatment with oral appliance
  Beck inventories (BDI)
Sustained attention | From the baseline evaluation to one year after the treatment with oral appliance
  Psychomotor Vigilance Test (PVT)
Cognition - Memory | From the baseline evaluation to one year after the treatment with oral appliance
  Digit Symbol Substitution Test (DSST)
Cognition - Learning strategies | From the baseline evaluation to one year after the treatment with oral appliance
  Rey Auditory-Verbal Learning Test (RAVLT)
Cognition - Immediate and late memories | From the baseline evaluation to one year after the treatment with oral appliance
  Wechsler Memory Scale (WMS)
Cognition - Processing speed ability | From the baseline evaluation to one year after the treatment with oral appliance
  Stroop Color Test
Cognition - Visual attention | From the baseline evaluation to one year after the treatment with oral appliance
  Trail Making Test - TMT
Quality of sleep | From the baseline evaluation to one year after the treatment with oral appliance
  Pittsburgh Sleep Quality Index (PSQI)
Quality of life | From the baseline evaluation to one year after the treatment with oral appliance
  Functional Outcomes of Sleep Questionnaire (FOSQ)
Stress | From the baseline evaluation to one year after the treatment with oral appliance
  Teste de Lipp
Metabolism | From the baseline evaluation to one year after the treatment with oral appliance
  Blood analysis of metabolism
Autonomic nervous system analysis | From the baseline evaluation to one year after the treatment with oral appliance
  Heart rate variability

CONTACTS AND LOCATIONS:
Locations (1):
- Associação Fundo de Incentivo à Pesquisa (AFIP), São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] de Godoy LBM, Sousa KMM, Palombini LO, Poyares D, Dal-Fabbro C, Guimaraes TM, Tufik S, Togeiro SM. Long term oral appliance therapy decreases stress symptoms in patients with upper airway resistance syndrome. J Clin Sleep Med. 2020 Nov 15;16(11):1857-1862. doi: 10.5664/jcsm.8698. PMID 32686643
- [Derived] Godoy LBM, Palombini L, Poyares D, Dal-Fabbro C, Guimaraes TM, Klichouvicz PC, Tufik S, Togeiro SM. Long-Term Oral Appliance Therapy Improves Daytime Function and Mood in Upper Airway Resistance Syndrome Patients. Sleep. 2017 Dec 1;40(12). doi: 10.1093/sleep/zsx175. PMID 29045745